CLINICAL TRIAL: NCT04862156
Title: Continued Access Protocol Study for the Use of the OrganOx Metra Normothermic Machine Perfusion Device in Human Liver Transplantation
Brief Title: WP02 Continued Access Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA agreed that WP02 CAP could be stopped. The OrganOx metra device was approved on December 9, 2021. The 105 planned CAP patients will be included in the Post-Approval study (NCT05526326).
Sponsor: OrganOx Ltd. (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP02
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Normothermic Machine Perfusion (NMP) (Experimental): Following the routine retrieval procedure of the liver, it will be placed on the OrganOx metra for Normothermic Machine Perfusion (NMP) for transport per the Investigational Plan and the Instructions for Use.
  Interventions: Device: Normothermic Machine Perfusion (NMP)

INTERVENTIONS:
Device: Normothermic Machine Perfusion (NMP) — Storage and transportation of the donated liver using the OrganOx metra device.
  Other Names: OrganOx metra device

SUMMARY:
The single-arm continued access phase will be used to collect additional effectiveness and safety data to support the objectives and outcomes of the original IDE pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or greater
* Subject is registered as an active recipient on the UNOS waiting list for liver transplantation
* Subject, or legally authorized representative, is able and willing to give informed consent and HIPAA authorization
* Subject is able and willing to comply with all study requirements

Exclusion Criteria:

* Subject requiring all of the following at the time of transplantation:

  1. Oxygen therapy via a ventilator/respirator
  2. Inotropic support
  3. Renal replacement therapy
* Subject has acute/fulminant liver failure (UNOS status 1A)
* Subject undergoing simultaneous transplantation of more than one organ (e.g., liver and kidney)
* Subject is pregnant (as confirmed by urine or serum pregnancy test) or nursing
* Concurrent enrollment in another clinical trial. Subjects enrolled in clinical trials or registries where only measurements and/or samples are taken (NO TEST DEVICE or TEST DRUG USED) are allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - Loyola University Chicago, Maywood, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normothermic Machine Perfusion (NMP)
Started | 19
Completed | 14
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Normothermic Machine Perfusion (NMP)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 31.8 (20.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Early Allograft Dysfunction (EAD)
Description: Severity of immediate graft injury as measured by early allograft dysfunction (EAD).
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP)
Number analyzed (Participants) | 19
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Normothermic Machine Perfusion (NMP)
All-Cause Mortality (participants affected / at risk) | 2/19
Serious Adverse Events (participants affected / at risk) | 19/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normothermic Machine Perfusion (NMP) (N=19)
Infection (Infections and infestations) | 3
Hepatic (Hepatobiliary disorders) | 6
Autoimmune (Immune system disorders) | 1
Cardiovacular (Cardiac disorders) | 4
Dermatologic (Skin and subcutaneous tissue disorders) | 1
Genitourinary (Renal and urinary disorders) | 6
Surgical Bleeding (Surgical and medical procedures) | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 4
Hematology (Blood and lymphatic system disorders) | 1
Neurology/Psychiatry (Psychiatric disorders) | 3

LIMITATIONS AND CAVEATS:
The study was terminated and the 19 subjects were included in the New Enrollment PAS study (NCT05526326)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT04862156/Prot_SAP_000.pdf